CLINICAL TRIAL: NCT00802607
Title: Procurement of Normal and Abnormal Bone, Dermis and Adipose Tissue for Establishment of Cell Cultures and Tissue Analysis
Brief Title: Collection of Tissue Specimens for Analysis and Establishment of Cell Cultures
Status: Terminated | Type: Observational
Why Stopped: Collaborating site, Children's Hospital, no longer able to provide connective tissues for this study.
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909046; 09-D-N046
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2010-10

CONDITIONS: Bone Diseases; Connective Tissue Diseases
Keywords: Bone Diseases; Connective Tissue Diseases
MeSH Terms: conditions — Bone Diseases; Connective Tissue Diseases

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will collect bone, cartilage, tendon, ligament, skin and fat tissue from patients undergoing surgery at Children's National Medical Center in Washington,

...

DETAILED DESCRIPTION:
Background:

It is now apparent that virtually every human post-natal tissue contains some type of stem/progenitor cell population that is responsible for tissue turnover and repair. Our previous studies have identified a subset of human bone marrow stromal cells (BMSCs) that is multi-potent and able to regenerate bone, cartilage, myelosupportive stroma and adipocytes, whereas stromal cells derived from human spleen (SpSCs) and thymus (TSCs) only form myelosupportive stroma. Recent studies suggest that human adipose-derived stromal cells (ASCs) may be similar to BMSCs, whereas stromal cells derived from human dermis (DSCs) have none of these properties (and serve as a negative control for most experiments in vitro and in vivo). How similar or dissimilar these different stromal cell populations are has yet to be determined. Molecular profiling is needed to compare these different populations and in order to elucidate the factors that control differentiation stromal cells into one cell type or another.

Objectives:

Surgical waste (bone with red marrow, dermis, and adipose tissues) from males and females of varying ages undergoing clinically indicated surgical procedures will be used to establish stromal cell cultures to study the molecular profile and differentiation capacity of the stromal cell populations from different tissues, and to further characterize the regulation of gene expression and protein synthesis in these stem/progenitors cells.

Eligibility:

Any patient who is undergoing clinically indicated surgery that entails removal of bone with red marrow, dermis and adipose tissue.

Design:

Normal surgical waste (bone with red marrow, dermis, and adipose) from procedures that are performed on males and females at Children's Hospital will be placed in nutrient medium (provided by NIDCR) and sent to the NIDCR for the establishment of cell culture strains. Only the age, gender, site from which the tissue was removed and clinical diagnosis will be recorded. The cell cultures from the different tissues will be used to determine their phenotypic character and differentiation properties by molecular profiling, and for studies to elucidate the regulation of gene expression and protein synthesis. Similarly, a portion of the samples obtained at Children's Hospital will be used to generate histological sections of the tissues. In some cases, RNA will be extracted from the tissues for RT-PCR analysis. Normal samples (cells, sections, mRNA) will also serve as normal controls for studies performed on samples obtained from patients with various diseases recruited to NIH under current NIH protocols (97-D-0055, 97-D-0145, 01-D-0184). Pathological samples (cells, sections, mRNA) will be studied in order to elucidate the cause of disease.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Any patient who is undergoing clinically indicated surgery that entails removal of bone with red marrow, dermis and adipose tissue.
* Patients with a documented musculoskeletal disease will be eligible for inclusion in this protocol if they are undergoing a medically indicated surgical procedure in which surgical waste containing bone and/or skin and/or fat is generated.
* Subjects under 18 years of age may be entered into this research study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-12-02 (Actual); Primary Completion 2010-10-04 (Actual); Study Completion 2010-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Bianco P, Riminucci M, Kuznetsov S, Robey PG. Multipotential cells in the bone marrow stroma: regulation in the context of organ physiology. Crit Rev Eukaryot Gene Expr. 1999;9(2):159-73. doi: 10.1615/critreveukargeneexpr.v9.i2.30. PMID 10445154
- [Background] Friedenstein AJ, Chailakhyan RK, Latsinik NV, Panasyuk AF, Keiliss-Borok IV. Stromal cells responsible for transferring the microenvironment of the hemopoietic tissues. Cloning in vitro and retransplantation in vivo. Transplantation. 1974 Apr;17(4):331-40. doi: 10.1097/00007890-197404000-00001. No abstract available. PMID 4150881
- [Background] Gronthos S, Franklin DM, Leddy HA, Robey PG, Storms RW, Gimble JM. Surface protein characterization of human adipose tissue-derived stromal cells. J Cell Physiol. 2001 Oct;189(1):54-63. doi: 10.1002/jcp.1138. PMID 11573204